CLINICAL TRIAL: NCT01329159
Title: Cardio-Respiratory Health in High Altitude Residents Exposed to Indoor Pollution
Brief Title: Cardio-Respiratory Health and Indoor Pollution
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Università degli Studi di Ferrara (Other)
Collaborators: Fondazione C.N.R./Regione Toscana "G. Monasterio", Pisa, Italy (Other Government)
Responsible Party: Annalisa Cogo, University of Ferrara
Other Study IDs: HA indoor/pollution
Record Dates: First submitted 2011-04-01; First posted 2011-04-05 (Estimated); Last update posted 2011-04-05 (Estimated); Status verified 2011-03

CONDITIONS: Pulmonary Disease; Cardiovascular Disease
Keywords: High altitude; respiratory function; cardiorespiratory health; indoor pollution
MeSH Terms: conditions — Lung Diseases; Cardiovascular Diseases; Altitude Sickness; Respiratory Aspiration

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to assess in the sample of population resident in the KHUMBU valley (NEPAL):

1. the respiratory function decline by means of spirometry and the respiratory health by means of questionnaire and six-minute walking distance
2. the presence of markers of early atherosclerosis with ultrasound and to estimate the value of systolic pulmonary pressure in comparison with not exposed subjects.

The investigators hypothesize that the chronic exposure to indoor pollution

1. can accelerate the physiological respiratory function decline, usually around 15-20mL/year in healthy subjects
2. induce cardiovascular impairment

   The population of high altitude villages is a unique sample to study the effect of the only indoor pollution. In fact, the absence of traffic, due to the lack of roads, and the very low level of smoking habits allow to have no other confounding factors
3. to study and analyze how the architectural features of the buildings of the village (distribution of domestic locals, natural or non natural ventilation systems, domestic activities, materials used, etc.) affect the indoor pollution from carbon monoxide, which necessarily is developed indoor during the daily life activities.

What the project prospects is to gather information focused on the scale of the building, independently from the typology, to study a model that will help to describe which aspects are most important to what concern the genesis of the pollution of the indoor air.

ELIGIBILITY:
Inclusion Criteria:

* residents in the villages of the valley

Exclusion Criteria:

* under the age of 14

Ages: 14 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: residents in the Kumbu Valley (Nepal)
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2011-04; Primary Completion 2012-04 (Estimated); Study Completion 2012-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Annalisa Cogo, MD, Study Director — University of Ferrara, Italy; Lorenza Pratali, MD, Principal Investigator — Institute of Clinical Physiology National Council of Research, Pisa, Italy; Luca Pomidori, PhD, Principal Investigator — Università degli Studi di Ferrara; Sanjay Nath Khanal, MD, Principal Investigator — Kathmandu University; Enrico Duo, Principal Investigator — Università degli Studi di Ferrara; Maria Rosa Bruno, MD, Principal Investigator — Institute of Clinical Physiology National Council of Research, Pisa, Italy; Chan Bahadur Thapa, MD, Principal Investigator — Tribhuvan University Institute of Medicine (Nepal)
Locations (1):
- Department of Clinical and Experimental Medicine- section of Respiratory Disease-University of Ferrara, Ferrara, Ferrara, Italy